CLINICAL TRIAL: NCT05595044
Title: Impact of Serum Vitamin D Correction on the Inflammatory Markers and Habilitation Outcome in Children With Autism Spectrum Disorder
Brief Title: Effect of Vitamin D Therapy in Autism Spectrum Disorder
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Mansour, Assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MansouraA
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Vitamin D; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Two study groups. One group receiving vitamin D plus habilitation and the other group receiving habilitation only
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D therapy and habilitation (Experimental): 40 ASD children receiving Vitamin D therapy and habilitation
  Interventions: Drug: Vitamin D; Other: Habilitation
- Habilitation (Other): 40 ASD children receiving habilitation
  Interventions: Other: Habilitation

INTERVENTIONS:
Drug: Vitamin D — ASD children with vitamin D insufficiency and deficiency will receive vitamin D with dose 300 IU/KG/ day not exceed 5000IU/day for 6 weeks then revaluate serum level of vitamin D if they reach normal level of vitamin D they will receive vitamin D 1000IU/ day till the end of 4 months.
  Arms: Vitamin D therapy and habilitation
Other: Habilitation — Habilitation

SUMMARY:
The aim of this work is to study the adjuvant effect of vitamin D supplementation on inflammatory marker (IL4) and habilitation outcome in children with Autism Spectrum Disorder in order to evaluate its efficiency as a treatment option based on correction of immune dysfunction.

DETAILED DESCRIPTION:
Vitamin D is one of environmental factors potentially modulating brain development and functioning. Vitamin D3 deﬁciency during pregnancy and early childhood is suggested to be one of several risk factors for development of ASD in genetically predisposed individuals (Cies´lin´ska et al., 2017). Many studies e.g (Eyles et al., 2013; Grant and Sole, 2009; Noriega and Savelkoul, 2014) suggested that vitamin D has an important role as a neuroactive steroid, which can affect neuronal differentiation, axonal connectivity and brain structure and function. Vitamin D has been increasingly recognized for its immunomodulatory role and has been implicated in the pathogenesis of autoimmune disorders. Also it has numerous and dynamic effects on the immune system, ranging from altering T cell responses and regulating cytokine pathways (Kocˇovská et al., 2017). So from this point of view, this study will be conducted to show adjuvant effect of vitamin D supplementation on ASD children at clinical level and inflammatory marker (IL4).

ELIGIBILITY:
Inclusion Criteria:

1. Delayed language development due to ASD.
2. Good nutritional status (Normal weight and height using growth charts, no Anemia and no clinical evidence of vitamin deficiency).
3. Normal hearing and vision.

Exclusion Criteria:

1. History of vitamin D supplementation, drugs modulating immune system as steroid and drug formula containing vitamin D as cod liver oil.
2. Known chronic disease.
3. Known neurological disorders or psychiatric disorders.
4. Known autoimmune or gastrointestinal disorders.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
language ability test | 4 months
  language test for assessment of language age
CARS questionnaire for assessment of ASD severity | 4 months
  CARS questionnaire for assessment of ASD severity
Inflammatory marker | 4 months
  Assessment of serum interleukin 4 by ELISA technique
Serum vitamin D | 6 weeks
  Assessment of serum vitamin D by ADVIA Centaur® Vitamin D Total (VitD) assay

CONTACTS AND LOCATIONS:
Overall Officials: Amira M. Mansour, MSc, Principal Investigator — Phoniatric unit, ORL department, faculty of medicine, Mansoura university
Locations (1):
- Mansoura university hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Vitamin D level, interleukin 4 in ASD
Supporting Information: Study Protocol, SAP
Time Frame: 2 years
Access Criteria: https://www.mans.edu.eg/